CLINICAL TRIAL: NCT00720551
Title: Calibration and Validation of the STISIM Driving Simulator: Simulated Driving Performance Under the Influence of Alcohol (0.05%, 0.08% AND 0.11%), and Placebo
Brief Title: Calibration and Validation of the STISIM Driving Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Responsible Party: Dr. J.C. Verster, Utrecht University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 07-374
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Simulated Driving Performance
Keywords: STISIM; Alcohol
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: alcohol — alcohol 0.05%, 0.08% or 0.11% or placebo

SUMMARY:
The aim of this study is to calibrate the STISIM driving simulator under influence of three different dosages of ethanol (0.05%, 0.08% and 0.11% BAC). The levels of performance decrement for the three blood alcohol concentrations will serve as a standard for comparing the effects that will be observed with psychoactive drugs in future trials. This will make the results of these future studies more easily to interpret and will provide health care providers and policy makers who read our scientific work with an easy-to-understand and clinically relevant comparison.

ELIGIBILITY:
Inclusion Criteria:

* 21-50 years old
* Written informed consent
* Normal static binocular acuity, corrected or uncorrected
* Normal hearing
* Social Drinker (average of 7 to 21 alcoholic drinks per week and experience with drinking 4-6 drinks per occasion)
* No current or past drug use
* Possession of a driver's license for at least 3 years
* Be considered as reliable and mentally capable of adhering to the protocol

Exclusion Criteria:

* Current and past drug use (positive urine drug screen on the presence of amphetamines (including MDMA), barbiturates, cannabinoids, benzodiazepines, cocaine, and opiates)
* Positive urine pregnancy screen in women
* Present use of psychoactive medication
* Positive alcohol breath test
* Prior enrollment in the same study
* Physical or mental illness
* Excessive alcohol use ( > 21 alcoholic drinks per week)
* Excessive smoking (more than 10 cigarettes per day)
* Intake of caffeine-containing beverages over 5 glasses per day
* Simulator sickness, as determined during the training session

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of the Lateral Position (SDLP) | one day

SECONDARY OUTCOMES:
Number of collisions and traffic violations | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joris C Verster, PhD, Principal Investigator — Utrecht University; Lieke M de Senerpont Domis, MSc, Study Director — Utrecht University
Locations (1):
- Utrecht University, Section Psychopharmacology, Utrecht, Netherlands

REFERENCES:
- [Derived] Mets MA, Kuipers E, de Senerpont Domis LM, Leenders M, Olivier B, Verster JC. Effects of alcohol on highway driving in the STISIM driving simulator. Hum Psychopharmacol. 2011 Aug;26(6):434-9. doi: 10.1002/hup.1226. Epub 2011 Aug 5. PMID 21823173